CLINICAL TRIAL: NCT06319469
Title: The Additive Value of Pyridostigmine to Silodosin in the Management of Acute Urinary Retention Secondary to Benign Prostatic Hyperplasia
Brief Title: The Additive Value of Pyridostigmine to Silodosin in Acute Urinary Retention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, ALshaimaa Ibrahim Rabie, principle investigator, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMBSUREC/06122022/Mohamed
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — silodosin; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group B (Experimental): 8 mg silodosin
  Interventions: Drug: silodosin 8 mg capsule
- group A (Experimental): silodosin 8 mg capsule and the pyridostigmine bromide 60 mg tablet
  Interventions: Drug: silodosin 8 mg capsule and the pyridostigmine bromide 60 mg tablet

INTERVENTIONS:
Drug: silodosin 8 mg capsule and the pyridostigmine bromide 60 mg tablet — The participants were assigned to groups A and B. Group B received the 8 mg silodosin capsule. In contrast, Group A was administered the silodosin 8 mg capsule and the pyridostigmine bromide 60 mg tablet. Over a week, each group administered their designated drug once per day
  Other Names: Siloprostat 8 mg and pyriclonerve 60 mg
  Arms: group A
Drug: silodosin 8 mg capsule — The participants were assigned to groups A and B. Group B received the 8 mg silodosin capsule. In contrast, Group A was administered the silodosin 8 mg capsule and the pyridostigmine bromide 60 mg tablet. Over a week, each group administered their designated drug once per day
  Other Names: Siloprostat 8 mg
  Arms: group B

SUMMARY:
Acute urine retention, AUR, is often considered the most serious consequence of aging men with progressive benign prostatic hyperplasia (BPH). AUR is defined as the sudden and painful inability to void freely. This study aims to evaluate whether pyridostigmine bromide added to silodosin is beneficial in treating acute urine retention caused by BPH.

DETAILED DESCRIPTION:
AUR, or acute urine retention, is often considered the most serious consequence of aging men with progressive benign prostatic hyperplasia (BPH). AUR is defined as the sudden and painful inability to void freely. (Hartung, 2001).

Between 0.4 and 25% of males seen in routine urological care are reported to have AUR each year (Schulman, 2001). According to a significant US cohort study, if a 60-year-old man survived for another 20 years, his probability of experiencing an AUR episode would be 23% (Jacobsen et al., 1997).

The current standard of care for AUR typically involves immediate bladder catheterization, followed by subsequent removal of the catheter to test whether normal voiding returns, that is, a trial without a catheter (TWOC) (Gwon et al., 2023).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a retention volume of less than 1000 milliliters who were over 50 years old and going through their first episode of acute urine retention (AUR) due to benign prostatic hyperplasia (BPH) were included in this study

Exclusion Criteria:

* The individuals who do not meet the eligibility requirements are those who have been diagnosed with an infection of the urinary tract, have repeatedly retained urine, have had unsuccessful trial voiding procedures in the past, have a retention volume of more than one liter, have had a history of prostatic or bladder neck surgery, have been diagnosed with prostate carcinoma, have experienced urethral stricture, have a neurogenic bladder, have been diagnosed with renal failure, or have been diagnosed with liver disease.

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 140 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
International Prostate Symptom Score (IPSS) | 3 MONTHS
  t is a validated, reproducible scoring system to assess disease severity and response to therapy. The IPSS is made up of 7 questions related to voiding symptoms. A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: ALSHAIMAA Ibrahim, Principal Investigator — BENISEUF UNIVERSITY
Locations (1):
- Beni-Seuf University Hospital, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: No
upon reasonable request